CLINICAL TRIAL: NCT00886977
Title: Pilot-Study of YAM80 in Amyotrophic Lateral Sclerosis. Evaluation of the Efficacy and Safety of YAM80 in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Efficacy and Safety of YAM80 in Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yoshino Neurology Clinic (Other)
Responsible Party: Hiide Yoshino, Clinic Director, Yoshino Neurology Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YAM80-01
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2009-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YAM80 — Oral administration, 2 to 6 mg, once a day.

SUMMARY:
The efficacy and safety are evaluated when YAM80 is administered orally to the patients of Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 25 and 65 years
* ALS patients who can visit the clinic for six months
* Forced Vital Capacity (FVC) > 70%
* Patients who can walk by themselves
* Change in ALSFRS-R score from -1 to -4 during 12 weeks before the initial administration
* Patients who are willing to give informed consent

Exclusion Criteria:

* Tracheotomy and invasive ventilation
* Pregnant or possibly pregnant female patients
* Female patients of childbearing potential who cannot practice contraception during and two years after the administration, and male patients who cannot practice contraception during and six months after the administration
* Patients with clinically significant conditions such as cardiovascular, respiratory, haematological, and renal diseases.
* Patients who are being treated with investigational drugs
* Patients who are treated with other ALS drugs within 2 weeks prior to the first administration

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R | 24w + follow-up period
Safety | 24w and the follow up period

SECONDARY OUTCOMES:
Manual Muscle Testing | 24w + follow-up period
Grip/pinch strength | 24w + followup period
Pulmonary function (forced vital capacity) | 24w + follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Hiide Yoshino, M.D., Principal Investigator — Yoshino Neurology Clinic
Locations (1):
- Yoshino Neurology Clinic, Tokyo, Japan